CLINICAL TRIAL: NCT04540770
Title: A Phase 1 Single and Multiple Dose Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Immunogenicity of HuL001 in Healthy Volunteers and Idiopathic Pulmonary Fibrosis Subjects
Brief Title: A Phase 1 Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Immunogenicity of HuL001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HuniLife Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: HuL001-CT-101
Record Dates: First submitted 2020-08-25; First posted 2020-09-07 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part A 1 (1 mg/kg HuL001) (Placebo Comparator): 6 healthy subjects will be enrolled and randomized to receive 1 dose of HuL001 (n = 4) or 1 dose of placebo (n = 2).
  Interventions: Drug: HuL001
- Part A 2 (3 mg/kg HuL001) (Placebo Comparator): 6 healthy subjects will be enrolled and randomized to receive 1 dose of HuL001 (n = 4) or 1 dose of placebo (n = 2).
  Interventions: Drug: HuL001
- Part A 3 (5 mg/kg HuL001) (Placebo Comparator): 6 healthy subjects will be enrolled and randomized to receive 1 dose of HuL001 (n = 4) or 1 dose of placebo (n = 2).
  Interventions: Drug: HuL001
- Part B 1 (Selected Dose) (Experimental): At the end of Part A, the SRC will review the accumulated unblinded data of safety, tolerability, PK (any available data), and immunogenicity (any available data) to select a dose to initiate Part B in IPF subjects. Part B will be conducted in multiple-dose, uncontrolled, and open-label manner to explore the safety, tolerability, PK, and immunogenicity in IPF subjects. Only one cohort will be enrolled to receive 3 repeated doses of the selected HuL001 dose, which will be administered bi-weekly.
  A total of 6 IPF subjects will be enrolled in this multiple-dose cohort.
  Interventions: Drug: HuL001

INTERVENTIONS:
Drug: HuL001 — Anti-ENO1 monoclonal antibody
  Other Names: Anti-Enolase 1 monoclonal antibody

SUMMARY:
This is a first-in-human, two-part, Phase 1 study that will characterize the safety, tolerability, PK, and immunogenicity of HuL001.

DETAILED DESCRIPTION:
This is a first-in-human, two-part, Phase 1 study that will characterize the safety, tolerability, PK, and immunogenicity of HuL001 after single ascending doses in healthy subjects followed by multiple doses in IPF subjects. The study will be conducted in 2 parts:

* Part A will enroll 3 single ascending doses (SAD) cohorts in healthy subjects. (HuL001:Placebo=4:2)
* Part B will enroll 1 multiple-dose cohort in IPF subjects. The proposed dose of HuL001 will be selected from the single-dose range of HuL001 evaluated in the healthy subjects of Part A. (HuL001=6)

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet the following criteria will be eligible to participate in the study:

Healthy and IPF Subjects

1. Female subjects and male subjects with female partners of child-bearing potential must agree to use adequate contraception (2 forms of birth control, one of which must be a barrier method). This criterion must be followed from the time of the first dose of treatment.
2. Able to understand, sign the written informed consent form, and follow the study procedures.
3. With no clinically significant abnormalities in vital signs, 12-lead ECG, and clinical laboratory assessments at screening as judged by the Investigator
4. Corrected QT interval using Fridericia's (QTcF) < 450 milliseconds (msec).

Healthy Subjects only

1. Aged between 20 and 55 years of age inclusive, at the time of signing the informed consent.
2. Alanine aminotransferase (ALT), alkaline phosphatase (ALP), and bilirubin ≤ 1.5x upper limit of normal (ULN) (isolated bilirubin > 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%).
3. Body weight ≥ 50 kilogram (kg), < 75 kg and body mass index (BMI) within the range 19.0 - 29.9 kg/m2 (inclusive).

IPF Subjects only

1. Aged between 40 and 90 years of age inclusive, at the time of signing the informed consent.
2. FVC≥ 40% and DLCO≥30%
3. Alanine aminotransferase (ALT), alkaline phosphatase (ALP), and bilirubin ≤ 2x upper limit of normal (ULN) (isolated bilirubin > 2xULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%).
4. Diagnosis of IPF as defined by ATS/ERS/JRS/ALAT guidelines (Raghu 2018) within the past 7 years prior to study participation.
5. Patients who are ineffective with an approved therapy (i.e., pirfenidone or nintedanib), or who are judged by the Investigator to be unsuitable for receiving approved therapy

Exclusion Criteria:

Subjects presenting with any of the following criteria will be excluded from participating in the study:

Healthy and IPF Subjects

1. Female subjects who are breastfeeding, pregnant, or planning to become pregnant during the study period.
2. The Investigator considers that the subject is not in the condition to participate in this study.
3. Evidence or history of clinically significant (as judged by the Investigator) hematologic, renal, endocrine, pulmonary (except for IPF subjects), gastrointestinal, cardiovascular (except for IPF subjects), hepatic, psychiatric, immunologic, metabolic, urologic, dermatologic, neurologic or allergic diseases, or other significant clinical findings within 3 months prior to screening.
4. Has participated in a clinical trial and has received an investigational product (IP) within 60 days prior to screening.
5. Previous history of anaphylaxis and severe allergic reaction, generation of neutralizing antibodies, or hypersensitivity to albumin or a protein-based therapeutic, or any other monoclonal antibody.
6. Had blood donation within 60 days or had blood donation over 250 mL within 90 days prior to screening, or cannot commit to stopping blood donation during the study period.
7. Receipt of vaccination within 1 month of screening or plan to receive vaccination during the study.
8. Have significant active infection (acute or chronic) within 28 days prior to screening.

Healthy Subjects only

1. A positive test for Human Immunodeficiency Virus (HIV) antibody, Hepatitis B surface antigen, or Hepatitis C antibody result within 3 months of screening.
2. Abnormal baseline blood tests exceeding any of the limits defined below:

   * ALT or aspartate transaminase (AST) > 1.5x ULN, ALP and bilirubin > 1.5x ULN (isolated bilirubin > 1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%)
   * Total white blood cell count < 2,500/mm3; subjects with lymphocyte count less than the Lower Limit of Normal (LLN) may be included at the Investigator's discretion; platelet count < 95,000/mm3
   * Creatinine > 2x ULN, calculated creatinine clearance < 60 mL/min (per Cockcroft & Gault)
   * International Normalized Ratio (INR) larger than upper limit of the normal reference range (0.9 - 1.3)
3. Current chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
4. Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 14 days or 5 half-lives (whichever is longer) prior to screening, unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise subject safety.
5. Previous exposure to any chimeric, humanized, or human monoclonal antibody, whether licensed or investigational.
6. Using tobacco products, nicotine products (patches, gum etc.) within 6 months prior to screening.

IPF Subjects only

1. A positive test for Human Immunodeficiency Virus (HIV) antibody, or Hepatitis C antibody result within 3 months of screening.
2. Abnormal baseline blood tests exceeding any of the limits defined below:

   * ALT or aspartate transaminase (AST) > 2x ULN, ALP and bilirubin > 2x ULN (isolated bilirubin > 2x ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%)
   * Total white blood cell count < 2,500/mm3; subjects with lymphocyte count less than the Lower Limit of Normal (LLN) may be included at the Investigator's discretion; platelet count < 95,000/mm3
   * Creatinine > 2x ULN, calculated creatinine clearance < 60 mL/min (per Cockcroft & Gault)
   * International Normalized Ratio (INR) larger than upper limit of the normal reference range (0.9 - 1.3)
3. Interstitial lung disease other than IPF.
4. Medical conditions, e.g., recent MI/stroke, severe chronic heart failure, pulmonary hypertension, or cancers, unsuitable for the study in the opinion of Investigator.
5. Acute IPF exacerbation during Screening.
6. Relevant airways obstruction (pre-bronchodilator FEV1/FVC< 0.7).
7. History of allergic or anaphylactic reaction to human, humanized, chimeric or murine monoclonal antibodies.
8. Treatment with prescription drugs for IPF within 5 half-lives of the drug, whichever is longer, prior to dosing.
9. Major surgery (major according to the investigator's assessment) planned during the course of the trial. (Being on a transplant list is allowed).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Frequency, severity, and causality of adverse events (AEs), including solicited local AEs | 70 Days in Part A and 84 Days in Part B
  Frequency, severity, and causality of adverse events (AEs), including solicited local AEs
Proportion of subjects who report clinically significant abnormal findings in physical examination | 70 Days in Part A and 84 Days in Part B
  Proportion of subjects who report clinically significant abnormal findings in physical examination
Change from baseline in blood pressure | 70 Days in Part A and 84 Days in Part B
  Change from baseline in systolic and diastolic blood pressure
Change from baseline in respiratory rate | 70 Days in Part A and 84 Days in Part B
  Change from baseline in respiratory rate
Change from baseline in heart rate | 70 Days in Part A and 84 Days in Part B
  Change from baseline in heart rate
Change from baseline in body temperature | 70 Days in Part A and 84 Days in Part B
  Change from baseline in body temperature
Change from baseline in hematology assessments | 70 Days in Part A and 84 Days in Part B
  The hematology assessments including hematocrit, hemoglobin, platelet count, red blood cell (RBC) count, white blood cell (WBC) count (total and differential), reticulocyte count and absolute neutrophil count.
Change from baseline in biochemistry assessments | 70 Days in Part A and 84 Days in Part B
  The biochemistry assessments including alanine aminotransferase (ALT), albumin, alkaline phosphatase (ALP), amylase, aspartate aminotransferase (AST), bicarbonate, blood urea nitrogen (BUN), calcium, chloride, creatinine, creatinine kinase, gamma glutamyl transferase (GGT), glucose, lactic acid dehydrogenase (LDH), lipid panel (low and high density lipids cholesterol, triglycerides; total cholesterol), magnesium, potassium, sodium, total bilirubin, total protein and uric acid.
Change from baseline in electrocardiogram (ECG) results (including PR, QRS, QT, QTcF, and RR intervals) | 70 Days in Part A and 84 Days in Part B
  Change from baseline in electrocardiogram (ECG) results
Tolerability of HuL001 in terms of frequency of events meeting the intra-cohort stopping criteria within the tolerability observation period | 70 Days in Part A and 84 Days in Part B
  Tolerability of HuL001 in terms of frequency of events meeting the intra-cohort stopping criteria within the tolerability observation period

SECONDARY OUTCOMES:
PK of single ascending doses of HuL001 in healthy subjects and multiple doses of HuL001 in IPF subjects- maximum observed concentration (Cmax) | 70 Days in Part A and 84 Days in Part B
  PK of single ascending doses of HuL001 in healthy subjects and multiple doses of HuL001 in IPF subjects- maximum observed concentration (Cmax)
PK of single ascending doses of HuL001 in healthy subjects and multiple doses of HuL001 in IPF subjects-time to reach Cmax (tmax) | 70 Days in Part A and 84 Days in Part B
  PK of single ascending doses of HuL001 in healthy subjects and multiple doses of HuL001 in IPF subjects-time to reach Cmax (tmax)
PK of single ascending doses of HuL001 in healthy subjects and multiple doses of HuL001 in IPF subjects- area under the curve from zero up to time t (AUC0-t) | 70 Days in Part A and 84 Days in Part B
  PK of single ascending doses of HuL001 in healthy subjects and multiple doses of HuL001 in IPF subjects- area under the curve from zero up to time t (AUC0-t)
PK of single ascending doses of HuL001 in healthy subjects and multiple doses of HuL001 in IPF subjects- apparent total clearance of the drug from plasma (CL/F) | 70 Days in Part A and 84 Days in Part B
  PK of single ascending doses of HuL001 in healthy subjects and multiple doses of HuL001 in IPF subjects- apparent total clearance of the drug from plasma (CL/F)
PK of single ascending doses of HuL001 in healthy subjects and multiple doses of HuL001 in IPF subjects- terminal half-life (t1/2) | 70 Days in Part A and 84 Days in Part B
  PK of single ascending doses of HuL001 in healthy subjects and multiple doses of HuL001 in IPF subjects- terminal half-life (t1/2)
PK of single ascending doses of HuL001 in healthy subjects and multiple doses of HuL001 in IPF subjects- apparent volume of distribution during terminal phase (Vz/F) | 70 Days in Part A and 84 Days in Part B
  PK of single ascending doses of HuL001 in healthy subjects and multiple doses of HuL001 in IPF subjects- apparent volume of distribution during terminal phase (Vz/F)
Proportion of subjects with positive anti-HuL001 antibodies | 70 Days in Part A and 84 Days in Part B
  Proportion of subjects with positive anti-HuL001 antibodies
Change from baseline in serum levels of cytokines | 70 Days in Part A and 84 Days in Part B
  Change from baseline in serum levels of cytokines

OTHER OUTCOMES:
Mean percent change from baseline of migrated PBMCs after single dose of HuL001 in healthy subjects (Cohort 1 of Part A only) and after the first and third doses of HuL001 administration in IPF subjects (Part B). | 0 Days in Part A and 0 Days,28 Days in Part B
  Mean percent change from baseline of migrated PBMCs after single dose of HuL001 in healthy subjects (Cohort 1 of Part A only) and after the first and third doses of HuL001 administration in IPF subjects (Part B).

CONTACTS AND LOCATIONS:
Overall Officials: Hao-Chien Wang, MD, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - Mackay Memorial Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No